CLINICAL TRIAL: NCT01051076
Title: Immune Tolerance Induction Study in Patients With Severe Type A Haemophilia With Inhibitor After Failure of a Previous Induction of Immune Tolerance With FVII Concentrates Without Von Willebrand Factor Rescue
Brief Title: Rescue Immunotolerance Study in Induction of Immune Tolerance (ITI)-Experienced Patients (RES.I.S.T. Experienced)
Acronym: RESIST EXP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: Charta Foundation (Other); Grifols Biologicals, LLC (Industry); CSL Behring (Industry); Biotest Pharmaceuticals Corporation (Industry); Grifols Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06200; 2008-007019-33 (EudraCT Number)
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Last update posted 2021-08-23 (Actual); Status verified 2020-12

CONDITIONS: Severe Hemophilia A
Keywords: ITI; Haemophilia A; Inhibitors; Failed ITI; VWF/FVIII concentrates
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII; optivate; factor VIII, von Willebrand factor drug combination; von Willebrand Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Factor VIII and von Willebrand Factor (Experimental)
  Interventions: Drug: VWF/FVIII concentrates

INTERVENTIONS:
Drug: VWF/FVIII concentrates — 200 IU/Kg by one or two bolus injections daily. After successful confirmation the dose will be tailed off progressively until discontinuation. Patients will be treated with a VWF/FVIII concentrates according to physician/patients preference.
  Other Names: Koate-DVI; Emoclot DI; Factane; 8Y; Optivate; Alphanate; Fahndi; Haemate P; Humate P; Haemoctine SDH; Octanate; Wilate

SUMMARY:
The purpose of this study is to evaluate whether a concentrate containing both FVIII and von Willebrand Factor (VWF) given at a high dose will induce immune tolerance in subjects who have already experienced and failed ITI with VWF-free FVIII concentrates. The treatment on this study is expected to last up to 33 months.

DETAILED DESCRIPTION:
The presence of Factor VIII (FVIII) inhibitor prevents FVIII infusions from working properly and makes treatment of bleeding episodes very difficult. Having an inhibitor is a serious and life-threatening complication in patients with Hemophilia. The usual treatment of patients with FVIII inhibitors involves what is called "immune tolerance induction" (ITI). Immune Tolerance means that the body can accept infused FVIII and that FVIII is again effective in controlling bleeds. ITI involves giving high doses of FVIII regularly until the inhibitor disappears. This treatment is not always effective. The inhibitor persists in about 1 in 5 patients who undergo ITI.

There are 2 types of FVIII concentrates: FVIII concentrates derived from human plasma, which contain VWF, and concentrates of FVIII without VWF. Both types of concentrates are commonly used to induce immune tolerance in patients with Hemophilia A. Retrospective studies on subjects who were treated with VWF containing Factor VIII concentrates after failing ITI with pure factor VIII concentrates, have shown that tolerance can be achieved in a large percentage of patients. This study will access prospectively whether treatment with a FVIII concentrate containing VWF given at a high dose (200 units per kilogram) daily for up to 33 months is able to induce immune tolerance after previous attempts with concentrates containing only FVIII have failed.

ELIGIBILITY:
Inclusion Criteria:

1. severe hemophilia A (FVIII<1%) with high responding inhibitors (peak levels >5 BU)
2. male, any age;
3. any inhibitor level at study enrollment;
4. ability and willingness to participate to the study;
5. previous ITI course of at least 9 months with a VWF-free FVIII concentrate at any dosage, such as recombinant FVIII and/or monoclonally purified FVIII.

Exclusion Criteria:

1. concomitant systemic treatment with immunosuppressive drugs;
2. concomitant experimental treatment;
3. previous history of myocardial infarction and/or cerebral stroke

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-11-03 (Actual); Primary Completion 2020-10-21 (Actual); Study Completion 2020-10-21 (Actual)

PRIMARY OUTCOMES:
Achievement of an inhibitor titer of <0.6 BU/failure to achieve an inhibitor titer of <0.6 BU within 33 months, or failure to decrease inhibitor titer by at least 20% compared to titer in prior 6 months, beginning at 3 months after starting ITI | 3 years
  Primary end point is the achievement of an inhibitor titer of less than 0.6 BU or failure to achieve an inhibitor titer of less than 0.6 BU within 33 months of treatment, or failure to decrease the inhibitor titer by at least 20% compared to the titer in the prior 6 months, beginning at 3 months after starting ITI

SECONDARY OUTCOMES:
Time to achieve success- either partial or complete. | 33 months
Safety - assessment of adverse events through treatment and compliance with prolonged regimen. | 33 months
  Includes assessment and evaluation of adverse events occurring through treatment and compliance with a lengthy regimen
Cost of care. | Up to 45 months
  Direct cost will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Nadia P. Ewing, MD, Principal Investigator — Clinical Professor of Pediatrics, City of Hope National Medical Center, Dept. of Pediatrics, 1500 E. Duarte Rd. Duarte, CA 91010
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

REFERENCES:
- [Background] Berntorp E, Ekman M, Gunnarsson M, Nilsson IM. Variation in factor VIII inhibitor reactivity with different commercial factor VIII preparations. Haemophilia. 1996 Apr;2(2):95-9. doi: 10.1111/j.1365-2516.1996.tb00022.x. PMID 27214015
- [Background] Kreuz W, Steiner J, Auerswald G, Beeg T, Becker S. Successful immunetolerance therapy of FVIII-inhibitor in chldren after changing from high to intermediate purity FVIII concentrate. Ann Hematol 1996; 72 (suppl 1).
- [Background] Gringeri A, Musso R, Mazzucconi MG, Piseddu G, Schiavoni M, Pignoloni P, Mannucci PM; RITS-FITNHES Study Group. Immune tolerance induction with a high purity von Willebrand factor/VIII complex concentrate in haemophilia A patients with inhibitors at high risk of a poor response. Haemophilia. 2007 Jul;13(4):373-9. doi: 10.1111/j.1365-2516.2007.01484.x. PMID 17610550
- See also: Related Info — http://www.isth.org
- See also: Related Info — http://www.wfh.org
- See also: Related Info — http://www.eahad.org
- See also: Related Info — http://www.hemophilia.org
- See also: Related Info — http://www.aiceonline.it